CLINICAL TRIAL: NCT06443476
Title: A Comparative Study Between Tenting Abutment Technique Versus Screw"Tent-Pole" Technique for Augmentation of Posterior Atrophic Mandible Randomized Clinical Trial
Brief Title: Tenting Abutment Technique Versus Screw"Tent-Pole" Technique for Augmentation of Posterior Atrophic Mandible
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohmmed Salem Hafedh, PRINCIPLE INVESTIGATOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS (3-3-5)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-06

CONDITIONS: Posterior Atrophic Mandible
Keywords: SANTA; tent abutment; Tent pole

STUDY DESIGN:
Intervention Model Description: Evaluate bone gained (height and width) and the period of time of healing in the atrophic posterior mandible when using the tenting abutment technique compared to the tent pole
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): Using a tent pole to gain bone in the atrophic posterior mandible.
  Interventions: Procedure: Tent pole technique
- study group (Active Comparator): Using a Tenting abutment to gain bone in the atrophic posterior mandible
  Interventions: Procedure: Tenting abutment technique

INTERVENTIONS:
Procedure: Tenting abutment technique — To evaluate a novel method using a designed tenting abutment to reduce number of surgeries and the edentulous healing period is shortened. In addition, to prevent vertical and horizontal collapse of the bone graft and minimizes resorption of the bone graft during the healing the atrophic posterior mandible.
  Arms: study group
Procedure: Tent pole technique — using the Tent pole technique to gain bone vertical and horizontal loss
  Arms: conventional group

SUMMARY:
To evaluate a novel method using a designed tenting abutment to reduce number of surgeries and the edentulous healing period is shortened. In addition, to prevent vertical and horizontal collapse of the bone graft and minimizes resorption of the bone graft during the healing the atrophic posterior mandible.

The tent pole provides excellent mechanical properties; stability & fixation, yet very poor features to preserve the integrity of the soft tissue.

Using the tenting abutment technique will help preserve the soft tissue and decrease the amount of dehiscence that might accompany the use of the tent pole.

DETAILED DESCRIPTION:
Augmentation of insufficient bone volume can be brought about by different methods, including, particulate and block grafting materials, guided Bone Regeneration with or without growth and differentiation factors, ridge splitting, expansion and distraction osteogenesis, either alone or in combination. These techniques may be used for horizontal/vertical ridge augmentation.

Xenograft bone has been utilized for the reconstruction of large 3-dimensional defects because it has no donor site morbidity and is of an unlimited volume in quantity.

Guided bone regeneration (GBR) describes the use of membranes to regenerate bony defects. A membrane for GBR needs to be biocompatible, cell occlusive, non-toxic, moldable and possess space-maintaining properties including stability.

* e. Explanation for choice of comparators (conventional titanium mesh): Tent pole offers superb mechanical properties for guided bone regeneration treatment in larger areas and it is regarded one of the most available covers for guided bone regeneration yet one of the cheapest.

  B. Objectives:
* a. Aim of the study:

  * To evaluate the quantity of gained bone under tenting abutment compared to a tent pole.
  * To evaluate amount of wound dehiscence postoperatively using tenting abutment technique compared to a tent pole.
  * ·To optimize the anatomical situation in order to facilitate implant installation.

7b. Hypothesis:

* Bone is a dynamic and living tissue with the capacity to repair and regenerate in response to injury. It is further possible to guide bone cells into an area that previously consisted of bony tissue to regenerate bone and increase the bone volume.
* Tenting abutment is suitable as a biomaterial for creating a space between the bone cortex and the periosteum to enhance new bone regeneration.
* Tenting abutment material will enhance the quantity and quality of newly formed bone.
* Tenting abutment will cause less soft tissue dehiscence and will dramatically decrease the percentage of the collapse of the space produced by the bone graft and minimizes resorption of the grafting material compared to the titanium mesh.

  7c. Primary and secondary objectives:
  1. Primary objective:

     Evaluate bone gained (height and width) and the period of time of healing in the atrophic posterior mandible when using tenting abutment technique compared to tent pole.
  2. Secondary objectives:

Evaluation of soft tissue dehiscence and resorption of the grafting material that might occur using tent pole compared to the tenting abutment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic posterior mandible.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicates implant placement

Exclusion Criteria:

* Local criteria:

  * Untreated gingivitis, periodontitis.
  * Insufficient oral hygiene.
  * Previous radiation therapy for the head and neck neoplasia, or bone augmentation to implant site..

Systemic criteria:

* Systemic disorders.
* Heavy smoking of more than 20 cigarettes per day.
* Bone pathology.
* ·Psychiatric problems. Emotional instability. Unrealistic aesthetic demands.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
height gained and width gained | before and post operative four months
  height gained and width gained Measure unit milimerter (mm) Measure device :CBCT

SECONDARY OUTCOMES:
Soft tissue dehiscence | after one month
  measure clinically (yes-no)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed ahmed Farid shehab, professor, Study Director — supervisor
Locations (1):
- Alaa Mohammed Hafedh, Cairo, Egypt